CLINICAL TRIAL: NCT01431170
Title: A Prospective, Double-Blinded, Parallel-Group, Randomized Study to Assess the Safety and Efficacy of Besivance™ for Treatment of Congenital Nasolacrimal Duct Obstruction in Children
Brief Title: Safety and Efficacy Study of Besivance™ for Treatment of Congenital Nasolacrimal Duct Obstruction in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0120110184
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-03

CONDITIONS: Congenital Nasolacrimal Duct Obstruction
MeSH Terms: interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Besivance Treatment Group (Experimental): Besivance™ ophthalmic suspension, 0.6%
  Interventions: Drug: Besivance Treatment Group
- Polytrim Treatment Group (Active Comparator): Polytrim ophthalmic solution
  Interventions: Drug: Polytrim Treatment Group

INTERVENTIONS:
Drug: Besivance Treatment Group — Subjects Receive Besivance™ ophthalmic suspension, 0.6% one drop in the study eye three times daily (TID) for 10 days.
  Other Names: Besifloxacin,Besivance
  Arms: Besivance Treatment Group
Drug: Polytrim Treatment Group — Subjects receive Polytrim ophthalmic solution one drop in the study eye three times daily (TID) for 10 days.
  Other Names: polymyxin b/trimethoprim - ophthalmic
  Arms: Polytrim Treatment Group

SUMMARY:
The goal of the study is to evaluate the application of Besivance™ (besifloxacin ophthalmic suspension, 0.6%) to treat congenital nasolacrimal duct obstruction in children. The hypothesis of the study is that Besivance™ is as safe and effective as the current standard of care for the treatment of nasolacrimal duct obstruction in children.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and efficacy of Besivance™ as an antibiotic treatment for congenital nasolacrimal duct obstruction with infection in children. The primary outcome measure is the change from baseline on the physician rated scale of Nasolacrimal Duct Obstruction (NLDO)with infection to follow-up visit #2 (Week 8) or at the time of treatment failure, if earlier.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have been diagnosed with congenital Nasolacrimal Duct Obstruction (NLDO) with infection by the Principal Investigator
* Both males and females
* Persons who are age of 1 to 12 months at time of diagnosis (time of diagnosis is defined as when the Principal Investigator makes clinical diagnosis.)

Exclusion Criteria:

* Persons who have received any antibiotic treatment for NLDO with infection for more than 2 week in the past 4 weeks.
* Persons who are currently receiving systemic antibiotic treatment that cannot be discontinued.
* Persons with any other ocular anomalies that could potentially interfere with interpretation of study results.
* Persons who have had any prior nasolacrimal duct system procedures such as stenting or probing.
* Persons who have previously participated in any clinical trial(s) of Besivance™
* Persons who have participated in any other clinical trial(s) of any investigational agent(s) within 30 days prior to the Baseline visit
* Persons who have any chronic diseases that might interfere with study participation

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suqin Guo, M.D., Principal Investigator — Institute of Ophthalmology and Visual Science, RUTGERS-New Jersey Medical School
Locations (1):
- Institute of Ophthalmology and Visual Science, RUTGERS-New Jersey Medical School, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Besivance Treatment Group: Subjects receive Besivance™ ophthalmic suspension, 0.6% one drop in the study eye three times daily for 10 days.
- Polytrim Treatment Group: Subjects receive Polytrim ophthalmic solution one drop in the study eye three times daily for 10 days.
Period: Overall Study
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Besivance Treatment Group: Subjects received Besivance™ ophthalmic suspension, 0.6% one drop in the study eye three times daily (TID) for 10 days.
- Polytrim Treatment Group: Subjects received Polytrim ophthalmic solution one drop in the study eye three times daily (TID) for 10 days.
- Total: Total of all reporting groups
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 110.83 (93.05) | 158.58 (110.62) | 134.71 (102.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Physician-rated Scale of NLDO From Baseline to Follow-Up Visit at Week 8 or From Baseline to Time of Treatment Failure, if Earlier.
Description: The NLDO grading scale in the study eye at every visit. The scale ranges from 0 to +4:
  * 0: No tearing and discharge.
  * 1: Tearing, moderate mucous discharge around nasolacrimal punctum
  * 2: Moderate redness of the medial eyelid with mucous discharge
  * 3: Redness and swelling of the eyelid with mucopurulent discharge
  * 4: Redness and swelling of eyelid with purulent discharge
  Due to varying baseline severity (measured by NLDO grade) among subjects, change from baseline to week 8 in NLDO grade was further classified as the following:
  Treatment success: grade of 0 or improvement by 2 or more compared to the prior visit.
  Recurrence: NLDO with infection returns in the study eye, as indicated by a NLDO grade >0 after a grade of 0 at the prior visit.
  Treatment Failure: grade is worse than or same as the baseline visit.
Time Frame: Baseline to Week 8
Measure: Number; unit: participants
Groups:
- Besivance Treatment Group: Subjects received Besivance ophthalmic solution in the study eye, one drop three times a day for ten days
- Polytrim Treatment Group: Subjects received Polytrim ophthalmic solution in the study eye, one drop three times daily for ten days.
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Number analyzed (Participants) | 9 | 11
participants
  Number of Treatment Success | 7 | 10
  Number of Recurrence | 1 | 1
  Number of Treatment Failure | 1 | 0

2. Secondary Outcome: Number of Recurrences by Randomization Group
Description: Recurrence is defined as when the NLDO with infection in the subject's study eye returns, as indicated by a NLDO grading scale of greater than zero after achieving a grade of zero at the previous visit.
  Number of subjects who had a recurrence event of the subjects who completed the study by treatment Group.
Time Frame: Baseline to Week 16 (Closeout Visit )
Population: The overall study recurrence rate was 10% study-wide (2 of 20 subjects), with one Besivance subject (11%), and one Polytrim subject (9%) experiencing recurrence.
Measure: Number; unit: Recurrence Subjects
Groups:
- Besivance Treatment Group: Number of subjects who had a recurrence randomized to the Besivance treatment group.
- Polytrim Treatment Group: Number of subjects who had a recurrence randomized to the Polytrim treatment group,
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Number analyzed (Participants) | 9 | 11
Recurrence Subjects | 1 | 1

3. Secondary Outcome: Efficacy of Recurrence Treatment as Measured by Change in the Physician- Rated Scale of NLDO
Description: Subjects who experience recurrence were re-treated as if they were a new patient, with the same study medication, were followed up then classified as "Treatment Success" or "Treatment Failure" according to study protocol.
Time Frame: Baseline to Week 16 (Closeout Visit)
Measure: Number; unit: participants
Groups:
- Efficacy of Besivance Treatment Group: Number of subjects who had a recurrence randomized to the Besivance treatment group.
- Efficacy of Polytrim Treatment Group: Number of subjects who had a recurrence randomized to the Polytrim treatment group,
Arm/Group | Efficacy of Besivance Treatment Group | Efficacy of Polytrim Treatment Group
Number analyzed (Participants) | 1 | 1
participants
  Number of Treatment Success after Recurrence | 1 | 0
  Number of Treatment Failure after Recurrence | 0 | 1

4. Secondary Outcome: Treatment Failure
Description: Possible treatment failure at a follow-up examination is operationally defined as follows: if the physician-grading scale of NLDO is worse than or same as the prior visit at any given follow-up visit, possible treatment failure then exists.
  Treatment Failure occurred if at visit #1 (2-week visit), the physician-grading scale of NLDO is worse than or same as the baseline visit. Treatment failure can also occur at recurrence visit #1 if the NLDO grading scale is worse or the same as compared to the previous visit. Subjects who meet the criteria for treatment failure were withdrawn from the study by the principal investigator and no additional data was collected. Subjects were referred for continued care.
Time Frame: Baseline to the time of failure or Week 16 (Closeout Visit)
Measure: Number; unit: Number of Treatment Failures
Groups:
- Besivance Treatment Group: Number of Treatment Failures for subjects randomized to the Besivance treatment group.
- Polytrim Treatment Group: Number of Treatment Failures for subjects randomized to the Polytrim treatment group.
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Number analyzed (Participants) | 9 | 11
Number of Treatment Failures | 1 | 1

5. Secondary Outcome: Medication Safety Outcomes
Description: During each study visit, the Principal Investigator will evaluate any possible adverse events by assessing clinical complaints and symptoms that are experienced by subjects and observed by the parent(s)/legal guardian(s), including findings in external, lacrimal duct system and anterior segment using slit lamp and fundus exam using indirect ophthalmoscope by principal investigator, as well as clinical signs including findings in external, nasolacrimal duct system and anterior segment using slit lamp and fundus exam using indirect ophthalmoscope by principal investigator.
Time Frame: Baseline to Week 16 (Closeout Visit )
Population: No safety issues were reported
Measure: Number; unit: Number of Adverse Events
Groups:
- Besivance Safety Outcomes: Number of reported medication safety issues in the Besivance Treatment Group.
- Polytrim Safety Outcomes: Number of reported medication safety issues in the Polytrim Treatment Group
Arm/Group | Besivance Safety Outcomes | Polytrim Safety Outcomes
Number analyzed (Participants) | 9 | 11
Number of Adverse Events | 0 | 0

6. Post Hoc Outcome: Number of Subjects Treated Successfully at Close-Out Visit (Week 16)
Description: Treatment Success is defined as a grade of 0 or improvement by 2 or more compared to the prior visit.
Time Frame: Baseline to Week 16 (Close-Out Visit)
Measure: Number; unit: Number of Treatment Success
Groups:
- Besivance Treatment Group: Number of subjects treated with Besivance™ ophthalmic suspension, 0.6%, who achieved treatment success by the study close-out visit (week 16).
- Polytrim Treatment Group: Number of subjects treated with Polytrim ophthalmic solution, who achieved treatment success by the study close-out visit (week 16).
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Number analyzed (Participants) | 9 | 11
Number of Treatment Success | 8 | 10

ADVERSE EVENTS:
Time Frame: Baseline to Closeout Visit (Week 16)
Groups:
- Besivance Treatment Group: Subjects randomized to the Besivance treatment group.
- Polytrim Treatment Group: Subjects randomized to the Polytrim treatment group.
Arm/Group | Besivance Treatment Group | Polytrim Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
Limitations include the small sample size which was reduced by participant drop out.We enrolled 24 subjects, completed and collected primary outcome measure data on 20.The recurrence rate was low at 10% (2 subjects), limiting secondary data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No